CLINICAL TRIAL: NCT00195377
Title: Evaluating Safety and QoL in Patients Treated With Etanercept: an Open Multicenter Study
Brief Title: Study Evaluating Etanercept in Patients With Rheumatoid Arthritis(RA), Juvenile Idiopathic Arthritis (JIA), or Psoriatic Arthritis (PsA) in Spain
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101393
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Arthritis, Psoriatic; Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to assess the safety of etanercept in patients with rheumatoid arthritis (RA), juvenile idiopathic arthritis (JIA) or psoriatic arthritis (PsA) in Spain

ELIGIBILITY:
Inclusion Criteria:

* RA or PsA in whom DMARDs/antiTNF antibodies/anti IL1 has been insufficient or inappropriate
* Children from 4 to 17 years old with JIA polyarticular

Exclusion Criteria:

* Clinically significant abnormal screening lab values
* Patients who are planning to undergo elective surgery during the study period.
* Other current autoimmune connective tissue diseases

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis, psoriatic arthritis or AIJ, treated with etanercept in rheumatology units
Sampling Method: Probability Sample
Enrollment: 1000
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Madrid, Madrid, Spain